CLINICAL TRIAL: NCT04052867
Title: Intravenous Lignocaine Infusion as a Multimodal Analgesic Approach in Laparoscopic Donor Nephrectomy
Brief Title: Intravenous Lignocaine Infusion in Laparoscopic Donor Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Consultant Anaesthesiologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: U1111-1237-9350
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain; Renal Transplantation; Morphine Adverse Reaction
Keywords: Intravenous lignocaine; Multimodal anagesic approach; Postoperative Pain; living related renal transplantation; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine group (Experimental): 20 patients undergoing elective laparoscopic donor nephrectomy will be given lignocaine infusion as part of the perioperative pain management.
  Interventions: Drug: Lignocaine
- Control group (Active Comparator): 20 patients undergoing elective laparoscopic donor nephrectomy will be receiving an equivalent volume of normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lignocaine — Slow bolus of lignocaine is given over 15 min before the start of surgery, followed by infusion of lignocaine
  Other Names: Intravenous lignocaine
  Arms: Lignocaine group
Drug: Normal saline — An equivalent volume of normal saline is given
  Arms: Control group

SUMMARY:
Background:

Administration of morphine as boluses or via a patient controlled analgesic device (PCA) has been the standard practice for donors after nephrectomy.

However, administration of morphine is far from being ideal analgesic as it does not provide optimal dynamic pain relief after major surgery, consistently demonstrate little effect on surgical stress response and organ dysfunction with high incidences of postoperative nausea/vomiting, respiratory depression and sedation. Several studies demonstrated perioperative intravenous lignocaine infusion can improve post-operative pain scores and morphine consumption in abdominal surgery.

The aim of this study is to identify the effectiveness of intra-operative lignocaine infusion in lowering postoperative pain and reduce postoperative morphine consumption in patients who undergo laparoscopic donor nephrectomy.

DETAILED DESCRIPTION:
Hypothesis:

Patients who receive intravenous lignocaine infusion as a multimodal analgesic technique will require less morphine postoperatively with lower pain scores on the visual analogue scale (VAS).

Methodology The main clinical study is a randomized double blinded control trial that will start after ethics approval from UMREC and registration at Clinical Trial Registry. All adults undergoing elective laparoscopic donor nephrectomy will be recruited in this double-blinded randomised controlled trial. After obtaining their informed consent, patients will be shown the visual analogue score (VAS) as the post-operative pain assessment and their baseline pain scores obtained. Instructions are also given for patient controlled analgesic (PCA) device using morphine for post-operative pain control.

Randomisation and blinding:

There will be two groups - lignocaine and control. Randomization will be based on a computer generated random number and sealed in opaque envelopes. On the day of surgery, one of the investigators who must not be involved in the care of the case, opens the envelope to follow the allocated group number and prepare either lignocaine or normal saline solutions. Both syringes are labelled with the assigned number only and handed to the attending anaesthesiologist in charge of the surgery. The patient as well as the attending anaesthetic team is blinded to the allocated group. Similarly, post-operative observers who collect the required data will be blinded.

Sample size:

Sample size is calculated based on a pilot study. A power analysis revealed that 15 patients in each group is required to detect a difference of 6 mg between the morphine consumption of the two groups for a power of 80% and and a level of statistical significance at 5%. To provide adequate power for additional analysis, we planned to enrol 20 patients in each group with further allowance for 10% drop out for the per protocol analysis.

Conduct of anaesthesia All patients are administered general anaesthesia with 2mcg/kg of fentanyl, 2-3mg/kg of propofol and 0.6mg/kg of rocuronium for induction, intubated and maintained with desflurane in oxygen-air mixture to MAC of 1.0-1.3. Haemodynamic parameters are measured with standard monitoring and kept within 10% of baseline. All management of ventilation, temperature control and fluids will be done according to institutional protocol for renal transplant.

Study drug protocol 2 groups - Control OR Lignocaine group. Lignocaine group: After induction, securing airway and intravenous lines, patients are turned lateral into the lateral decubitus nephrectomy position. Once the correct position is achieved and haemodynamic status is stable, a slow bolus of 1.5mg/kg of 1% lignocaine is given over 15 min before the start of surgery, followed by an infusion at 1.5mg/kg/hr for the lignocaine group. If the patient's BMI is >30, the ideal body weight (IBW) is used to calculate the bolus and infusion dose at a maximal rate of 100mg/hr for a wide margin of safety.

Control group: An equivalent volume of normal saline is given.

Multimodal analgesia All patients will receive

* 0.05-0.1 mg/kg of intravenous morphine intra-operatively.
* One gram of intravenous paracetamol and 40mg of intravenous parecoxib (30min before end of surgery) unless contraindicated.
* Anti-emetics - dexamethasone 4mg and IV ondansetron 4mg
* 20-30 mls of plain bupivacaine 0.5% (not exceeding 2mg/kg) will be infiltrated subcutaneously

In the recovery room, the PCA device is set to deliver 1mg bolus of morphine without a baseline infusion, lockout period of 5 min and maximum of 30mg morphine in 4 hours.

* The time to first PCA use is noted.
* Pain scores using VAS will be recorded at 30 min, 1 hour, 6 hours, 12 hours and 24 hours post-operatively.
* Other symptoms such as sedation, nausea, vomiting, light headedness, perioral numbness, and pruritus are reported if it occurs during the first postoperative day.

In the ward, oral paracetamol 1g 6hourly and oral celecoxib 200mg 12hourly will be prescribed for administration in the ward. Total IV morphine consumption at the end of the 24 hours are recorded.

Demographic data, medical history, physical examination, pre- and postoperative laboratory results for renal function (eGFR and creatinine clearance) will be collected prospectively. All post-operative pain scores/ satisfaction scores/ complications will be reviewed and recorded by a blinded observer.

4 blood samples will be taken from every recruited patient - baseline pre-op, before nephrectomy, after nephrectomy and 24 hours post-op.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic donor nephrectomy

Exclusion Criteria:

* refuse consent
* allergic to local anaesthetics or opioids,
* on long term analgesics for chronic pain,
* have impaired liver function
* has history of arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine requirement | 24 hours postoperatively
  Morphine usage post-operatively

SECONDARY OUTCOMES:
Level of systemic lignocaine | before lignocaine infusion, after lignocaine infusion just before nephrectomy, half hour after nephrectomy, within 24 post operatively
  Serial venous blood are taken at 4 different intervals

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, MBBS, MMed, Principal Investigator — University Malaya, Malaysia
Locations (1):
- University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathuram Thiyagarajan U, Bagul A, Nicholson ML. Pain management in laparoscopic donor nephrectomy: a review. Pain Res Treat. 2012;2012:201852. doi: 10.1155/2012/201852. Epub 2012 Oct 23. PMID 23150820
- [Background] Waller JR, Hiley AL, Mullin EJ, Veitch PS, Nicholson ML. Living kidney donation: a comparison of laparoscopic and conventional open operations. Postgrad Med J. 2002 Mar;78(917):153-7. doi: 10.1136/pmj.78.917.153. PMID 11884697
- [Background] Gerbershagen HJ, Dagtekin O, Rothe T, Heidenreich A, Gerbershagen K, Sabatowski R, Petzke F, Ozgur E. Risk factors for acute and chronic postoperative pain in patients with benign and malignant renal disease after nephrectomy. Eur J Pain. 2009 Sep;13(8):853-60. doi: 10.1016/j.ejpain.2008.10.001. Epub 2008 Nov 14. PMID 19010073
- [Background] Dolin SJ, Cashman JN, Bland JM. Effectiveness of acute postoperative pain management: I. Evidence from published data. Br J Anaesth. 2002 Sep;89(3):409-23. PMID 12402719
- [Background] Weibel S, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Afshari A, Kranke P. Efficacy and safety of intravenous lidocaine for postoperative analgesia and recovery after surgery: a systematic review with trial sequential analysis. Br J Anaesth. 2016 Jun;116(6):770-83. doi: 10.1093/bja/aew101. PMID 27199310
- [Background] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681
- [Background] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177